CLINICAL TRIAL: NCT06741111
Title: A Real-world Assessment in Implementation of the MASH Patient Care Pathway in Chinese Population Using the Meinian Health Check-up Database
Acronym: IMPACT MASH
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-8256; U1111-1308-1064 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-12-16; First posted 2024-12-18 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD) & Steatohepatitis (MASH)
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: People who underwent health check-up in Meinian check-up centres between the period January 1st, 2023, to December 31st, 2023
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The primary objective of this study is to estimate the proportion of people with low/intermediate/high risk of advanced fibrosis in at risk Chinese population based on the European Association for the Study of the Liver (EASL) 2024 care pathway

ELIGIBILITY:
Inclusion Criteria:

For All and Study population:

1. Male or female, age above or equal to 18 years on health-check-up visit day
2. No missing value on sex

For EASL at risk population

1. Must be part of study population.
2. People with T2D or [obesity＋above or equal to 1 cardiometabolic risk factor(s)] or elevated liver enzymes

For EASL not at-risk population

1. Must be part of study population.

For EASL-SAFE

1. Must be part of EASL at risk population

For AGA at risk population

1. Must be part of study population.
2. People with 2 or more metabolic risk factors (EASL-MASLD criteria) or T2D or steatosis on any imaging modality or with elevated aminotransferases

For CSH MAFLD population

1. Must be part of study population.
2. Liver steatosis on abdominal ultrasound
3. With at least one component of Metabolic syndrome (MetS [CSH])

Exclusion Criteria:

1. Individuals originating from centers with fewer than 100 participants
2. Missing value of liver stiffness measurement (LSM)
3. Had an interquartile range/median ratio above or equal to 30% of the measurement of LSM
4. Missing value on either aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or platelet count (PLT)
5. Missing value on FPG, TG, HDLc or BP (to define the presence of metabolic risk factors)
6. Missing value on abdominal ultrasound

For EASL not at-risk population 1. People with T2D or [obesity＋above or equal to 1 cardiometabolic risk factor(s)] or elevated liver enzymes

For EASL-SAFE/NFS

1. Missing value on globulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who underwent health check-up in Meinian check-up centres between January 1st, 2023 to December 31st, 2023 and met the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1233970 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
The proportion of people with low/intermediate/high risk of advanced fibrosis in EASL at risk population based on EASL 2024 care pathway. | January 1st, 2023, to December 31st, 2023
  Number and proportion of people in respective risk population

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bangalore, India

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com